CLINICAL TRIAL: NCT07316413
Title: Repetitive Transcranial Magnetic Stimulation in Frontotemporal Lobar Degeneration
Acronym: FTLD_rTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Barbara Borroni, Professor, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FTLD_rTMS
Record Dates: First submitted 2025-12-01; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-04

CONDITIONS: FTLD; FTD; bvFTD; PPA; PSP; Cortical Basal Syndrome (CBS); rTMS; Theta Burst Stimulation
MeSH Terms: conditions — Frontotemporal Lobar Degeneration

STUDY DESIGN:
Intervention Model Description: The study is structured in two phases. In the first phase, double-blind, randomised and placebo-controlled, participants will be randomised into two groups: group 1, participants will receive real rTMS for 2 weeks; and group 2, placebo rTMS for 2 weeks. In the second, open-label phase, after 10 weeks, both group 1 and group 2 participants will receive real rTMS for 2 weeks. Each participant will receive a total of 4 weeks of intervention (4 weeks of real stimulation in group 1, or 2 weeks of real stimulation and 2 weeks of placebo stimulation in group 2), with 5 sessions per week (Monday to Friday) lasting approximately 30 minutes each.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real iTBS - Real iTBS (Experimental): 10 sessions of theta burst stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of theta burst stimulation (5 days/week for 2 weeks)
  Interventions: Device: Theta burst stimulation
- Sham iTBS - Real iTBS (Sham Comparator): 10 sessions of sham stimulation (5 days/week for 2 weeks) followed by an open-label 10 sessions of theta burst stimulation (5 days/week for 2 weeks)
  Interventions: Device: Theta burst stimulation; Device: Sham Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — 10 sessions (5 days/week for 2 weeks) of 20 trains of 10 bursts, each containing 3 pulses at 50 Hz, applied at a frequency of 5 Hz (total pulses: 600, total duration: approx. 3 minutes); this protocol will be repeated twice within each single session.
Device: Sham Theta burst stimulation — 10 sessions (5 days/week for 2 weeks) of sham theta burst stimulation.The device providing Theta Burst Stimulation can be placed in the same position and turned on, creating a similar experience for the participant, without providing any neural stimulation.
  Arms: Sham iTBS - Real iTBS

SUMMARY:
The aim of the study is to evaluate the safety, feasibility, clinical and biological efficacy, and predictors of efficacy of an intervention consisting of repetitive transcranial magnetic stimulation (rTMS) in patients with frontotemporal dementia (FTLD) or in asymptomatic persons at risk of FTLD (i.e., persons familiar with FTLD patients).

rTMS is a non-invasive brain stimulation technique, and has demonstrated the ability to modulate neuronal activity by applying high-frequency magnetic fields to the surface of the skull. rTMS offers a potentially effective means to influence neural networks involved in the pathogenesis of neurodegenerative diseases, with benefits that could extend beyond symptomatic relief. Its safety has been widely documented in a variety of clinical conditions, making it an ideal candidate for application in neurodegenerative diseases.

In the present study, participants will undergo the following procedures: (i) clinical and neuropsychological assessment, (ii) TMS, and (iii) blood sampling. The occurrence of adverse events will be monitored throughout the duration of the study.

The study is structured in two phases. In the first phase, double-blind, randomised and placebo-controlled, participants will be randomised into two groups: group 1, participants will receive real rTMS for 2 weeks; and group 2, placebo rTMS for 2 weeks. In the second, open-label phase, after 10 weeks, both group 1 and group 2 participants will receive real rTMS for 2 weeks. Each participant will receive a total of 4 weeks of intervention (4 weeks of real stimulation in group 1, or 2 weeks of real stimulation and 2 weeks of placebo stimulation in group 2), with 5 sessions per week (Monday to Friday) lasting approximately 30 minutes each.

Visits will take place at the beginning of the study (T00) and after 2 weeks (T02, end of the first phase), 12 weeks (T12, beginning of the second phase), 14 weeks (T14, end of the second phase), 24 weeks (T24, follow-up). During each visit, participants underwent the following procedures: (i) clinical and neuropsychological assessment, (ii) blood sampling, and (iii) TMS. Specific biomarker analyses will be performed on the blood samples to study the pathophysiological mechanisms of the disease and the effect of the experimental intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of FTLD (bvFTD, avPPA, svPPA, CBS, or PSP)
* global CDR plus NACC FTLD ≤ 1

Exclusion Criteria:

* presence of cerebrovascular disease, hydrocephalus, intracranial masses identified by MRI, history of head trauma, serious medical conditions unrelated to FTLD, history of epilepsy, and presence of electronic (e.g., pacemaker) or metallic implants in the head.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety of repetitive Transcranial Magnetic Stimulation Protocol | Through study completion, at week 24
  Safety will be assessed in terms of the frequency and severity of any adverse events. Safety will be monitored throughout the duration of the study.
Feasibility of repetitive Transcranial Magnetic Stimulation Protocol | Through study completion, at week 24
  Feasibility will be assessed according to the study drop-out rate. Feasibility will be monitored throughout the duration of the study.
Effectiveness in restoring neurotransmission | Through study completion, at week 24
  Neurotransmission will be assessed by measuring changes in glutamatergic (intracortical facilitation, ICF) and GABAergic (short-interval intracortical inhibition, SICI) neurotransmission assessed indirectly through TMS.

SECONDARY OUTCOMES:
Clinical effectiveness | Change from baseline to week 2, 12, 14, 24
  Clinical effectiveness will be assessed by measuring changes in clinical and cognitive measures, in behavioural and neuropsychiatric symptoms, and in caregiver burden. Specifically, the following instruments will be used: Clinical Global Impression (CGI) Severity (CGI-S) and Improvement (CGI-I) and FBI.
Biological efficacy | Change from baseline to week 2, 12, 14, 24
  Biological efficacy will be assessed via blood sampling by measuring changes in neurodegeneration biomarkers: neurofilament light (NfL, measured in pg/mL); astrogliosis: Serum Glial Fibrillary Acidic Protein (GFAP, measured in pg/mL).
Predictors of efficacy | Change from baseline to week 2, 12, 14, 24
  We will assess whether demographic characteristics (age, gender, level of education), genetic traits (comparing genetic and sporadic forms of FTD), clinical phenotype (bvFTD, avPPA, svPPA, CBS, or PSP), disease severity, markers of cognitive reserve, and plasma biomarker profile are correlated with better treatment response.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Centro San Giovanni Di Dio - Fatebenefratelli Brescia, Brescia, Italy, Italy

REFERENCES:
- [Background] Antczak J, Kowalska K, Klimkowicz-Mrowiec A, Wach B, Kasprzyk K, Banach M, Rzeznicka-Brzegowy K, Kubica J, Slowik A. Repetitive transcranial magnetic stimulation for the treatment of cognitive impairment in frontotemporal dementia: an open-label pilot study. Neuropsychiatr Dis Treat. 2018 Mar 13;14:749-755. doi: 10.2147/NDT.S153213. eCollection 2018. PMID 29559782
- [Background] Dong K, Zhu X, Xiao W, Gan C, Luo Y, Jiang M, Liu H, Chen X. Comparative efficacy of transcranial magnetic stimulation on different targets in Parkinson's disease: A Bayesian network meta-analysis. Front Aging Neurosci. 2023 Jan 4;14:1073310. doi: 10.3389/fnagi.2022.1073310. eCollection 2022. PMID 36688161
- [Background] Wei Z, Fu J, Liang H, Liu M, Ye X, Zhong P. The therapeutic efficacy of transcranial magnetic stimulation in managing Alzheimer's disease: A systemic review and meta-analysis. Front Aging Neurosci. 2022 Sep 6;14:980998. doi: 10.3389/fnagi.2022.980998. eCollection 2022. PMID 36147701
- [Background] Siebner HR, Funke K, Aberra AS, Antal A, Bestmann S, Chen R, Classen J, Davare M, Di Lazzaro V, Fox PT, Hallett M, Karabanov AN, Kesselheim J, Beck MM, Koch G, Liebetanz D, Meunier S, Miniussi C, Paulus W, Peterchev AV, Popa T, Ridding MC, Thielscher A, Ziemann U, Rothwell JC, Ugawa Y. Transcranial magnetic stimulation of the brain: What is stimulated? - A consensus and critical position paper. Clin Neurophysiol. 2022 Aug;140:59-97. doi: 10.1016/j.clinph.2022.04.022. Epub 2022 May 18. PMID 35738037
- [Background] Menardi A, Rossi S, Koch G, Hampel H, Vergallo A, Nitsche MA, Stern Y, Borroni B, Cappa SF, Cotelli M, Ruffini G, El-Fakhri G, Rossini PM, Dickerson B, Antal A, Babiloni C, Lefaucheur JP, Dubois B, Deco G, Ziemann U, Pascual-Leone A, Santarnecchi E. Toward noninvasive brain stimulation 2.0 in Alzheimer's disease. Ageing Res Rev. 2022 Mar;75:101555. doi: 10.1016/j.arr.2021.101555. Epub 2021 Dec 30. PMID 34973457
- [Background] Benussi A, Alberici A, Samra K, Russell LL, Greaves CV, Bocchetta M, Ducharme S, Finger E, Fumagalli G, Galimberti D, Jiskoot LC, Le Ber I, Masellis M, Nacmias B, Rowe JB, Sanchez-Valle R, Seelaar H, Synofzik M; GENFI Consortium; Rohrer JD, Borroni B. Conceptual framework for the definition of preclinical and prodromal frontotemporal dementia. Alzheimers Dement. 2022 Jul;18(7):1408-1423. doi: 10.1002/alz.12485. Epub 2021 Dec 7. PMID 34874596
- [Background] Hoglinger GU, Respondek G, Stamelou M, Kurz C, Josephs KA, Lang AE, Mollenhauer B, Muller U, Nilsson C, Whitwell JL, Arzberger T, Englund E, Gelpi E, Giese A, Irwin DJ, Meissner WG, Pantelyat A, Rajput A, van Swieten JC, Troakes C, Antonini A, Bhatia KP, Bordelon Y, Compta Y, Corvol JC, Colosimo C, Dickson DW, Dodel R, Ferguson L, Grossman M, Kassubek J, Krismer F, Levin J, Lorenzl S, Morris HR, Nestor P, Oertel WH, Poewe W, Rabinovici G, Rowe JB, Schellenberg GD, Seppi K, van Eimeren T, Wenning GK, Boxer AL, Golbe LI, Litvan I; Movement Disorder Society-endorsed PSP Study Group. Clinical diagnosis of progressive supranuclear palsy: The movement disorder society criteria. Mov Disord. 2017 Jun;32(6):853-864. doi: 10.1002/mds.26987. Epub 2017 May 3. PMID 28467028
- [Background] Armstrong MJ, Litvan I, Lang AE, Bak TH, Bhatia KP, Borroni B, Boxer AL, Dickson DW, Grossman M, Hallett M, Josephs KA, Kertesz A, Lee SE, Miller BL, Reich SG, Riley DE, Tolosa E, Troster AI, Vidailhet M, Weiner WJ. Criteria for the diagnosis of corticobasal degeneration. Neurology. 2013 Jan 29;80(5):496-503. doi: 10.1212/WNL.0b013e31827f0fd1. PMID 23359374
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Rascovsky K, Hodges JR, Knopman D, Mendez MF, Kramer JH, Neuhaus J, van Swieten JC, Seelaar H, Dopper EG, Onyike CU, Hillis AE, Josephs KA, Boeve BF, Kertesz A, Seeley WW, Rankin KP, Johnson JK, Gorno-Tempini ML, Rosen H, Prioleau-Latham CE, Lee A, Kipps CM, Lillo P, Piguet O, Rohrer JD, Rossor MN, Warren JD, Fox NC, Galasko D, Salmon DP, Black SE, Mesulam M, Weintraub S, Dickerson BC, Diehl-Schmid J, Pasquier F, Deramecourt V, Lebert F, Pijnenburg Y, Chow TW, Manes F, Grafman J, Cappa SF, Freedman M, Grossman M, Miller BL. Sensitivity of revised diagnostic criteria for the behavioural variant of frontotemporal dementia. Brain. 2011 Sep;134(Pt 9):2456-77. doi: 10.1093/brain/awr179. Epub 2011 Aug 2. PMID 21810890
- [Background] Grossman M, Seeley WW, Boxer AL, Hillis AE, Knopman DS, Ljubenov PA, Miller B, Piguet O, Rademakers R, Whitwell JL, Zetterberg H, van Swieten JC. Frontotemporal lobar degeneration. Nat Rev Dis Primers. 2023 Aug 10;9(1):40. doi: 10.1038/s41572-023-00447-0. PMID 37563165
- [Background] Stokes MG, Chambers CD, Gould IC, Henderson TR, Janko NE, Allen NB, Mattingley JB. Simple metric for scaling motor threshold based on scalp-cortex distance: application to studies using transcranial magnetic stimulation. J Neurophysiol. 2005 Dec;94(6):4520-7. doi: 10.1152/jn.00067.2005. Epub 2005 Aug 31. PMID 16135552
- [Background] Taylor JJ, Newberger NG, Stern AP, Phillips A, Feifel D, Betensky RA, Press DZ. Seizure risk with repetitive TMS: Survey results from over a half-million treatment sessions. Brain Stimul. 2021 Jul-Aug;14(4):965-973. doi: 10.1016/j.brs.2021.05.012. Epub 2021 Jun 13. PMID 34133991
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Vacas SM, Stella F, Loureiro JC, Simoes do Couto F, Oliveira-Maia AJ, Forlenza OV. Noninvasive brain stimulation for behavioural and psychological symptoms of dementia: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2019 Sep;34(9):1336-1345. doi: 10.1002/gps.5003. Epub 2018 Oct 17. PMID 30246461
- [Background] Fox MD, Halko MA, Eldaief MC, Pascual-Leone A. Measuring and manipulating brain connectivity with resting state functional connectivity magnetic resonance imaging (fcMRI) and transcranial magnetic stimulation (TMS). Neuroimage. 2012 Oct 1;62(4):2232-43. doi: 10.1016/j.neuroimage.2012.03.035. Epub 2012 Mar 19. PMID 22465297